CLINICAL TRIAL: NCT06173856
Title: Effectiveness of Phototherapy With and Without Probiotics for the Treatment of Indirect Hyperbilirubinemia in Preterm Neonates
Brief Title: Effectiveness of Phototherapy With and Without Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Medical University (Other)
Responsible Party: Principal Investigator, Naeem Afzal, Professor, Fatima Jinnah Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAU-1
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy group (Active Comparator): LED phototherapy (430-470nm)
  Interventions: Other: LED phototherapy
- phototherapy with probiotics group (Experimental): In group B, LED phototherapy (430-470nm) with probiotics (125mg Saccharomyces boulardii, twice a day, orally mixed in 5cc of milk whichever the neonate is taking).
  Interventions: Other: LED phototherapy

INTERVENTIONS:
Other: LED phototherapy — LED phototherapy (430-470nm) alone will be applied.

SUMMARY:
Raised serum bilirubin levels can cause kernicterus and premature infants are at increased risk due to metabolic immaturity. The standard treatment for neonatal jaundice is phototherapy but probiotics along with it can reduce the duration of phototherapy and hospitalization stay, secondarily can reduce the risk of nosocomial infection.

DETAILED DESCRIPTION:
Raised serum bilirubin levels can cause kernicterus and premature infants are at increased risk due to metabolic immaturity. The comparative analytical study was conducted after the ethical approval for one year (Jan 2022-Jan 2023) in the neonatal unit of The University of Lahore Teaching Hospital, Lahore, Pakistan. 76 preterm neonates fulfilling the selection criteria were included in the study and divided into two groups.

Standard phototherapy was applied in both groups and group A probiotic (Saccharomyces boulardii) 125mg, twice daily, orally (in 5cc of milk whichever the baby was taking) was given till discharge from the hospital. The primary outcome measurements were the duration of phototherapy and the length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* All the Neonates with indirect hyperbilirubinemia,
* Born at ;37 weeks of gestation
* Both male and female neonates were included in the study

Exclusion Criteria:

* Neonates with sepsis,
* bilirubin level in exchange transfusion range
* direct hyperbilirubinemia
* Neonates with respiratory distress syndrome, severe birth asphyxia, intubated and critically sick

Ages: 0 Hours to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
effectiveness | 1 to 2 weeks
  mean duration of phototherapy and the mean duration of hospital stay with and without probiotics for treatment of indirect hyerbilirubinemia in preterm neonates probiotics for the treatment of indirect hyperbilirubinemia in preterm neonates

CONTACTS AND LOCATIONS:
Locations (1):
- Humaira Waseem, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No
when results are compiled